CLINICAL TRIAL: NCT02565628
Title: A Phase 1b, Double Blind, Sponsor Open, Randomized, Parallel, Group Multiple Dose Study Examining The Safety, Tolerability, Pharmacokinetics And Pharmacodynamics Of Pf-06669571 In Subjects With Idiopathic Parkinson's Disease.
Brief Title: PF-06669571 In Subjects With Idiopathic Parkinson's Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: B7821002
Record Dates: First submitted 2015-09-28; First posted 2015-10-01 (Estimated); Results first posted 2017-08-07 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2017-04

CONDITIONS: Idiopathic Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — PF-06669571

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- PF-06669571 (Experimental): Once daily (QD) for 7 days
  Interventions: Drug: PF-06669571
- Placebo (Placebo Comparator): QD for 7 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PF-06669571 — 1 milligram (mg) QD for 3 days followed by 3 mg QD for 4 days
  Arms: PF-06669571
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This study is designed to assess safety, tolerability and pharmacokinetic data for multiple doses of PF-06669571 in subjects with idiopathic Parkinson's disease. In addition, this study will assess whether PF-06669571 is able to demonstrate superior efficacy compared with placebo in the treatment of the motor symptoms of idiopathic Parkinson's disease.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have a clinical diagnosis of idiopathic Parkinson's disease and presence of at least 2 out of 3 cardinal characteristics (tremor, rigidity and/or bradykinesia).
* Must be Hoehn & Yahr Stage II-III inclusive and experiencing motor fluctuations in the form of end-of-dose wearing off during the morning hours or early morning akinesia.
* Subjects should be able to recognize their "wearing off" symptoms and verify that they usually improve after their next dose of Parkinson's disease medication. Subjects should be able to recognize drug-induced dyskinesias and verify whether or not they are troublesome.

Exclusion Criteria:

- History or clinical features consistent with an atypical parkinsonian syndrome, (for example: ataxia, dystonia, clinically significant orthostatic hypotension.

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-11-16 (Actual); Primary Completion 2016-05-13 (Actual); Study Completion 2016-05-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (9):
- United States (9):
  - Pfizer New Haven Clinical Research Unit, New Haven, Connecticut
  - MD Clinical, Hallandale, Florida
  - QPS-MRA, LLC (Broward Research Group), Hollywood, Florida
  - Qps-Mra Llc, South Miami, Florida
  - QPS-MRA, LLC (Miami research Associates), South Miami, Florida
  - QPS-MRA, LLC (MRA Clinical Research), South Miami, Florida
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - CRI Worldwide, LLC, Marlton, New Jersey
  - CTI Clinical Research Center, Cincinnati, Ohio

REFERENCES:
- [Derived] Gurrell R, Duvvuri S, Sun P, DeMartinis N. A Phase I Study of the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of the Novel Dopamine D1 Receptor Partial Agonist, PF-06669571, in Subjects with Idiopathic Parkinson's Disease. Clin Drug Investig. 2018 Jun;38(6):509-517. doi: 10.1007/s40261-018-0632-6. PMID 29478239
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B7821002&StudyName=A%20Phase%201b%2C%20Double%20Blind%2C%20Sponsor%20Open%2C%20Randomized%2C%20Parallel%2C%20Group%20Multiple%20Dose%20Study%20Examining%20The%20Safety%2C%20Tolerability%2C%20Pharmacokinetics%20And%20Pharmacodynamics%20Of%20Pf-06669571%20In%20Subjects%20With%20Idiopathic%20Parkinson%27s%20Disease.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 20 participants were randomized, 19 participants were treated. One participant was randomized but withdrew consent before receiving any treatment. This subject was not included in any analysis set.
Groups:
- PF-06669571 0.5 mg: PF-06669571 0.5 mg was orally administered on Day 1 through Day 7 as tablets. Participants swallowed 2 tablets on Days 1-3 (1 mg total) and 6 tablets (3 mg total) on Days 4-7 once daily, with ambient temperature water to a total volume of approximately 240 mL. A follow-up visit of 7-14 days after last dose of the treatment was completed.
- Placebo: Placebo matched to PF-06669571 was orally administered on Day 1 through Day 7 as tablets. Participants swallowed 6 tablets everyday with ambient temperature water to a total volume of approximately 240 mL. A follow-up visit of 7-14 days after last dose of the treatment was completed.
Period: Overall Study
Arm/Group | PF-06669571 0.5 mg | Placebo
Started | 10 | 9
Received Treatment | 10 | 9
Completed | 10 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PF-06669571 0.5 mg | Placebo | Total
Number analyzed (Participants) | 10 | 9 | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.5 (7.4) | 67.9 (5.9) | 66.6 (6.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 9
  Male | 6 | 4 | 10

OUTCOME MEASURES:

1. Primary Outcome: Maximum Percent Change From Baseline in Movement Disorder Society-Sponsor Revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Part III at Day 7.
Description: The total MDS-UPDRS score is the most common method of evaluating the severity of Parkinson's disease across behaviors, activities of daily living, motor abilities, and other complications of Parkinson's disease. The MDS-UPDRS focuses primarily on measuring impairments associated with Parkinson's disease, with subsections organized according to motor and non-motor aspects of the disease. Part III assesses the motor signs of Parkinson's disease. Higher total scores indicate more severe motor signs of Parkinson's disease. Negative changes from baseline indicate improvement. MDS-UPDRS Part III total motor score is comprised of 33 sub-scores based on 18 items, several with right, left or other body distribution scores. Each question is anchored with five responses that are linked to commonly accepted clinical terms: 0 = normal, 1 = slight, 2 = mild, 3 = moderate and 4 = severe.
Time Frame: Day 7
Population: All enrolled participants who started treatment.
Measure: Least Squares Mean (Standard Error); unit: Percentage
Arm/Group | PF-06669571 0.5 mg | Placebo
Number analyzed (Participants) | 10 | 9
Percentage | -19.24 (7.21) | -14.21 (7.60)
Statistical Analysis 1: Comparison: PF-06669571 0.5 mg vs Placebo; Test type: Superiority or Other; p = 0.6382, Mixed Models Analysis; Least Square Mean Difference = -5.02, 90% CI 1-sided [upper limit 8.97], Standard Error of Mean 10.49

2. Primary Outcome: Number of Participants in Each Columbia Classification Algorithm of Suicide Assessment (C-CASA) Category by Study Visit on Day -2, Day 8 or Early Withdrawal, and Early Withdrawal/Follow-Up Visit
Description: The number of participants in each C-CASA category was mapped from Columbia-Suicide Severity Rating Scale (C-SSRS) data. C-SSRS assessed whether participant experienced following: completed suicide (1), suicide attempt (2) (response of "Yes" on "actual attempt"), preparatory acts toward imminent suicidal behavior (3) ("Yes" on "preparatory acts or behavior"), suicidal ideation (4) ("Yes" on "wish to be dead", "non-specific active suicidal thoughts", "active suicidal ideation with methods without intent to act or some intent to act or some intent to act, with specific plan and intent"), any suicidal behavior or ideation, self-injurious behavior (7) ("Yes" on "Has subject engaged in non-suicidal self-injurious behavior").
Time Frame: Day -2, Day 8, and follow-up visit (Day 7 - 14 after last dose of PF-06669571)
Population: All enrolled participants who started treatment.
Measure: Number; unit: participants
Arm/Group | PF-06669571 0.5 mg | Placebo
Number analyzed (Participants) | 10 | 9
participants
  Day -2 | 0 | 0
  Day 8 | 0 | 0
  Follow-up visit | 0 | 0

3. Primary Outcome: Number of Participants With New Onset and Worsening of Post-Baseline Suicidality.
Description: Number of participants with new onset and worsening of post-baseline suicidality was reported
Time Frame: Day 8 or follow-up visit (Day 7 - 14 after last dose of PF-06669571)
Population: All enrolled participants who started treatment
Measure: Number; unit: participants
Arm/Group | PF-06669571 0.5 mg | Placebo
Number analyzed (Participants) | 10 | 9
participants | 0 | 0

4. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (All Causalities)
Description: An adverse event (AE) was any untoward medical occurrence in a clinical investigation subject administered a product or medical device; the event need not necessarily have a causal relationship with the treatment or usage.
Time Frame: Day 1 to 28 calendar days after the last dose of investigational product
Population: All enrolled participants who started treatment
Measure: Number; unit: participants
Arm/Group | PF-06669571 0.5 mg | Placebo
Number analyzed (Participants) | 10 | 9
participants | 6 | 5

5. Primary Outcome: Number of Participants With Supine and Standing Vital Sign Abnormalities of Potential Clinical Concern (Absolute Values)
Description: Number of participants with supine and standing vital signs data of absolute values meeting criteria of potential clinical concern. Absolute values were analyzed for supine/standing systolic blood pressure (SBP), supine/standing diastolic blood pressure (DBP), and supine/standing pulse rate. Number of participants with vital signs data meeting the following criteria was reported: (1) absolute supine SBP <90 millimeters of mercury (mmHg); (2) absolute standing SBP <90 mmHg; (3)absolute supine DBP<50mmHg; (4)absolute standing DBP<50mmHg (5) absolute supine pulse rate <40 beats per minute (bpm); (6) absolute supine pulse rate >120 bpm;(7) absolute standing pulse rate <40 bpm; (8) absolute standing pulse rate >140 bpm.
Time Frame: Screening, Days -1, 1, 7 and 8, and follow-up visit
Population: All enrolled participants who started treatment
Measure: Number; unit: participants
Arm/Group | PF-06669571 0.5 mg | Placebo
Number analyzed (Participants) | 10 | 9
participants
  Supine Systolic BP <90 mmHg | 0 | 0
  Standing Systolic BP <90 mmHg | 1 | 0
  Supine Diastolic BP <50 mmHg | 0 | 0
  Standing Diastolic BP <50 mmHg | 0 | 0
  Supine Pulse Rate <40 BPM | 0 | 0
  Supine Pulse Rate >120 BPM | 0 | 0
  Standing Pulse Rate <40 BPM | 0 | 0
  Standing Pulse Rate >140 BPM | 0 | 0

6. Primary Outcome: Number of Participants With Supine and Standing Vital Sign Abnormalities of Potential Clinical Concern (Increase From Baseline)
Description: The number of participants with vital signs data of maximum increase from baseline meeting the following criteria was reported: Criterion A: maximum increase from baseline in supine systolic BP (SBP) >=30 millimeters of mercury (mmHg); Criterion B maximum increase from baseline in standing SBP >=30 mmHg; Criterion C: maximum increase from baseline in supine diastolic BP(DBP) >=20 mmHg; Criterion D: maximum increase from baseline in standing diastolic BP(DBP) >=20 mmHg
Time Frame: Screening, Days -1, 1, 7 and 8, and follow-up visit
Population: All enrolled participants who started treatment
Measure: Number; unit: participants
Arm/Group | PF-06669571 0.5 mg | Placebo
Number analyzed (Participants) | 10 | 9
participants
  Criterion A | 1 | 1
  Criterion B | 0 | 1
  Criterion C | 0 | 1
  Criterion D | 1 | 1

7. Primary Outcome: Number of Participants With Supine and Standing Vital Sign Abnormalities (Decrease From Baseline)
Description: The number of participants with vital signs data of maximum decrease from baseline meeting the following criteria was reported: Criterion A: maximum decrease from baseline in supine systolic BP (SBP) >=30 mmHg; Criterion B: maximum decrease from baseline in standing SBP >=30 mmHg; Criterion C: maximum decrease from baseline in supine diastolic BP(DBP) >=20 mmHg; Criterion D: maximum decrease from baseline in standing diastolic BP(DBP) >=20 mmHg
Time Frame: Screening, Days -1, 1, 7 and 8, and follow-up visit
Population: All enrolled participants who started treatment
Measure: Number; unit: participants
Arm/Group | PF-06669571 0.5 mg | Placebo
Number analyzed (Participants) | 10 | 9
participants
  Criterion A | 5 | 3
  Criterion B | 4 | 2
  Criterion C | 3 | 3
  Criterion D | 3 | 2

8. Primary Outcome: Number of Participants With Electrocardiogram (ECG) That Met Categorical Criteria for Concern (Absolute Value)
Description: The number of participants with ECG absolute values meeting the following criteria was reported: Criterion A: maximum PR interval (time from the beginning of P wave to the start of QRS complex, corresponding to the end of atrial depolarization and onset of ventricular depolarization) >=300 msec; Criterion B: maximum QRs complex(time from Q wave to the end of S wave, corresponding to ventricle depolarization) >=140 msec; Criterion C: maximum QTcF interval (time from the beginning of Q wave to the end of T wave corresponding to electrical systole, corrected for heart rate using Fridericia's formula) 450-<480 msec; Criterion D: maximum QTcF interval 480-<500 msec; Criterion E: maximum QTcF interval (Fridericia's correction) >=500 msec
Time Frame: Screening, Days 1, 7, and 8, and follow-up visit
Population: All enrolled participants who started treatment
Measure: Number; unit: participants
Arm/Group | PF-06669571 0.5 mg | Placebo
Number analyzed (Participants) | 10 | 9
participants
  Criterion A | 0 | 0
  Criterion B | 0 | 0
  Criterion C | 0 | 0
  Criterion D | 0 | 0
  Criterion E | 0 | 0

9. Primary Outcome: Primary: Number of Participants With Electrocardiogram (ECG) That Met Categorical Criteria for Concern(Increase From Baseline)
Description: Number of participants with ECG(standard 12-lead) meeting the following criteria was reported: Criterion A: maximum PR interval increase from baseline percentage change (PctChg)>=25/50%; Criterion B: maximum QRs complex increase from baseline PctChg >=50%; Criterion C: maximum QTcF interval increase from baseline 30<=change<60 msec; Criterion D: maximum QTcF interval increase from baseline change >=60 msec.
Time Frame: Screening, Days 1, 7, and 8, and follow-up visit
Population: All enrolled participants who started treatment
Measure: Number; unit: participants
Arm/Group | PF-06669571 0.5 mg | Placebo
Number analyzed (Participants) | 10 | 9
participants
  Criterion A | 0 | 0
  Criterion B | 0 | 0
  Criterion C | 2 | 0
  Criterion D | 0 | 0

10. Primary Outcome: Number of Participants With Laboratory Abnormalities That Met Categorical Criteria for Concern (Without Regard to Baseline Abnormality)
Description: Number of participants with a laboratory abnormality meeting specified criteria. The laboratory test included: hematology (hemoglobin, hematocrit, red blood cell count, mean corpuscular volume, mean corpuscular hemoglobin, mean corpuscular hemoglobin concentration, platelet count, white blood cell count, absolute total neutrophils, absolute eosinophils, absolute basophils, absolute monocytes, and absolute lymphocytes),liver function(total bilirubin, direct bilirubin, aspartate, aspartate aminotransferase, alanine, alanine aminotransferase, alkaline phosphatase, total protein, and albumin), renal function (blood urea nitrogen, creatinine, and uric acid), electrolytes (sodium, potassium, chloride, calcium, and venous bicarbonate), clinical chemistry(glucose) ,and urinalysis (pH, qualitative glucose, qualitative protein, qualitative blood, qualitative ketones, qualitative bilirubin, nitrites, leukocyte esterase, urine urobilinogen, urine leukocyte, esterase and microscopy).
Time Frame: Screening, Days 1, 4, and 7, and follow-up visit
Population: All enrolled participants who started treatment.
Measure: Number; unit: participants
Arm/Group | PF-06669571 0.5 mg | Placebo
Number analyzed (Participants) | 10 | 9
participants | 8 | 5

11. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of PF-06669571 on Day 1 and Day 7
Description: Cmax of PF-06669671 was observed directly from data on Day 1 and Day 7
Time Frame: 0, 1, 3, 5, 8 and 12 hours post-dose on both Day 1 and Day 7
Population: The PF-06669571 pharmacokinetics(PK) concentration analysis set was used for this analysis, and it was defined as all subjects randomized and treated who have at least 1 measureable concentration of interest.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | PF-06669571 0.5 mg
Number analyzed (Participants) | 10
ng/mL
  Day 1 | 16.87 (30)
  Day 7 | 92.51 (31)

12. Secondary Outcome: Area Under Curve From Time Zero to 12 Hours (AUC12) of PF-06669571 on Day 1 and Day 7
Description: AUC12 of PF-06669571 refers to the area under the curve from time zero to 12 hours post dose on Day 1 and Day 7. AUC12 was determined by using linear/log trapezoidal method.
Time Frame: 0, 1, 3, 5, 8 and 12 hours post-dose on both Day 1 and Day 7
Population: The PF-06669571 PK parameter analysis set was used for this analysis, and it was defined as all subjects randomized and treated who have at least 1 of the PK parameters of interest measured.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | PF-06669571 0.5 mg
Number analyzed (Participants) | 10
ng*hr/mL
  Day 1 | 150.8 (28)
  Day 7 | 917.5 (35)

13. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) of PF-06669571 on Day 1 and Day 7
Description: Tmax of PF-06669571 was observed directly from data on Day 1 and Day 7, as time of first occurrence.
Time Frame: 0, 1, 3, 5, 8 and 12 hours post-dose on both Day 1 and Day 7
Population: The PF-06669571 PK concentration analysis set was used for this analysis, and it was defined as all subjects randomized and treated who have at least 1 measureable concentration of interest.
Measure: Mean (Full Range); unit: hr
Arm/Group | PF-06669571 0.5 mg
Number analyzed (Participants) | 10
hr
  Day 1 | 3.35 [1.40 to 8.42]
  Day 7 | 3.19 [1.42 to 5.42]

14. Secondary Outcome: Area Under Curve From Time Zero to 24 Hours (AUC24) of PF-06669571 on Day 7
Description: AUC24 of PF-06669571 refers to the area under the curve from time zero to 24 hours post dose on Day 7. AUC24 was determined by using linear/log trapezoidal method
Time Frame: 0, 1, 3, 5, 8, 12 and 24 hours post-dose on Day 7
Population: as for outcome 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | PF-06669571 0.5 mg
Number analyzed (Participants) | 10
ng*hr/mL | 1626 (38)

ADVERSE EVENTS:
Arm/Group | PF-06669571 0.5 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/9
Other Adverse Events (participants affected / at risk) | 6/10 | 5/9
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PF-06669571 0.5 mg (N=10) | Placebo (N=9)
Dry mouth (Gastrointestinal disorders) | 2 | 1
Nausea (Gastrointestinal disorders) | 2 | 2
Vomiting (Gastrointestinal disorders) | 1 | 2
Ill-defined disorder (General disorders) | 2 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0
Dystonia (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 1 | 0
Resting tremor (Nervous system disorders) | 0 | 1
Abnormal dreams (Psychiatric disorders) | 1 | 0
Nocturia (Renal and urinary disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.